CLINICAL TRIAL: NCT05844982
Title: A Trial Evaluating Intravitreal Faricimab (6.0 mg) Injections or Fluocinolone Acetonide (0.19 mg Intravitreal Implants vs Observation for Prevention of Visual Acuity Loss Due to Radiation Retinopathy
Brief Title: Intravitreal Faricimab Injections or Fluocinolone Acetonide (0.19 mg) Intravitreal Implants vs Observation for Prevention of VA Loss Due to Radiation Retinopathy
Acronym: AL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); National Institutes of Health (NIH) (NIH); Alimera Sciences (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Protocol AL; UG1EY014231 (NIH)
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Radiation Retinopathy; Visual Impairment
Keywords: Visual Acuity; Radiation retinopathy; Faricima; Fluocinolone Acetonide
MeSH Terms: conditions — Vision Disorders | interventions — faricimab; Fluocinolone Acetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intravitreal faricimab (Active Comparator): Study eyes assigned to receive faricimab will receive a dose of 6.0 mg of faricimab. Faricimab is supplied in a single use vial.
  Interventions: Drug: Faricimab
- Fluocinolone Acetonide Intravitreal Implants (Active Comparator): Study eyes assigned to receive fluocinolone acetonide intravitreal implant will receive a dose of 0.19 mg fluocinolone acetonide intravitreal implant (Iluvien). The implant is supplied in a sterile single use applicator with a 25-gauge needle
  Interventions: Drug: fluocinolone acetonide
- Observation (No Intervention)

INTERVENTIONS:
Drug: Faricimab — 6.0 mg intravitreal injection at randomization and every 3 months
  Arms: Intravitreal faricimab
Drug: fluocinolone acetonide — 0.19 mg fluocinolone acetonide intravitreal implant (Iluvien) at randomization and at 24 months
  Arms: Fluocinolone Acetonide Intravitreal Implants

SUMMARY:
This randomized controlled trial will evaluate the effect of intravitreal faricimab or fluocinolone acetonide (FAc) intravitreal implant compared with observation on long-term visual acuity following treatment of choroidal melanoma with iodine-125 plaque brachytherapy.

DETAILED DESCRIPTION:
The primary objectives are to compare long-term visual acuity outcomes in eyes that receive repeated treatment with faricimab or fluocinolone acetonide intravitreal implants with those observed initially and treated only if macular edema (ME) develops. The secondary objectives are to determine if repeated treatment with faricimab or fluocinolone acetonide intravitreal implants versus observation can prevent or alter the course of ME from radiation retinopathy and to evaluate the natural history of radiation retinopathy with multimodal imaging including widefield color photographs, widefield fluorescein angiography and OCTA.

ELIGIBILITY:
Key Inclusion Criteria

* Primary uveal melanoma (excluding iris melanoma) receiving primary treatment with plaque brachytherapy
* Absence of unrelated cause of visual loss
* Baseline visual acuity ≥ 34 letters (20/200 Snellen equivalent or better)
* Posterior tumor margin >0 mm from the center of the macula (i.e., tumor is NOT under the geometric center of the fovea)
* Posterior tumor margin >0 mm from the closest disc margin (i.e., tumor is not touching the edge of the optic disc)
* Calculated total dose to center of the macula ≥30 Gy

Key Exclusion Criteria

* Opaque media
* Inability to undergo fluorescein angiography
* Less than 18 years of age
* Prior vitrectomy
* Intraocular pressure (IOP) ≥ 25 mmHg or history of steroid- induced IOP elevation that required treatment at baseline
* IOP ≥ 25 mmHg at randomization or increase in IOP ≥ 8 mmHg from baseline to randomization (following steroid challenge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2029-12-26 (Estimated); Study Completion 2029-12-26 (Estimated)

PRIMARY OUTCOMES:
Change in visual acuity from baseline | from baseline at 3 years
  Visual acuity is measured as a continuous integer letter score from 0 to 100, with higher numbers indicating better visual acuity. A letter score of 85 is approximately 20/20 and a letter score of 70 is approximately 20/40, the legal unrestricted driving limit in most states. A 5-letter change for an individual is approximately equal to a 1-line change on a vision chart.
Loss of 15 or more letters of visual acuity from baseline | from baseline at 3 years
  Visual acuity is measured as a continuous integer letter score from 0 to 100, with higher numbers indicating better visual acuity. A letter score of 85 is approximately 20/20 and a letter score of 70 is approximately 20/40, the legal unrestricted driving limit in most states. A 5-letter change for an individual is approximately equal to a 1-line change on a vision chart.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - Retina Consultants, Manchester, Connecticut
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Northwestern Memorial Group, Chicago, Illinois
  - IL Eye and Ear Infirmary-University of Illinois at Chicago, Chicago, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - University of Iowa Department of Ophthalmology and Visual Sciences, Iowa City, Iowa
  - Foundation for Vision Research and Retina Specialists of Michigan, P.C., Grand Rapids, Michigan
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Retina Research Institute, LLC, St Louis, Missouri
  - The Cleveland Clinic Foundation DBA Cleveland Clinic Lerner College of Medicine, Celveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Retina-Vitreous Consultants, Inc., Monroeville, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Pittsburgh Clinical Trial Consortium, Sewickley, Pennsylvania
  - Retina Consultants of Carolina, PA, Greenville, South Carolina
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Consultants of Texas, PA, Bellaire, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Retina Associates, Lubbock, Texas
  - The Board of Regents of the University of Wisconsin System, Madison, Wisconsin